CLINICAL TRIAL: NCT04981535
Title: The Comparison of Level of Aerosol Particle at the Face Level of Endoscopist Performing Upper Gastrointestinal Endoscopy in Patients With and Without Head Box; a Randomized Control Trial
Brief Title: Aerosol Particle From EGD in Patients With and Without Head Box in COVID-19 Era
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Associate Professor, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP022
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: EGD; Covid19; Aerosol Disease; Head Box
Keywords: Upper gastrointestinal endoscopy; EGD; COVID-19; Aerosol-generating procedure; Head box
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing upper gastrointestinal endoscopy with head box (Experimental): experimental group
  Interventions: Device: Head box during upper gastrointestinal endoscopy
- Patients undergoing upper gastrointestinal endoscopy without head box (No Intervention): standard of care group

INTERVENTIONS:
Device: Head box during upper gastrointestinal endoscopy — "็Head box" is an acrylic box over a patient's head who undergoing upper gastrointestinal endoscopy.
  Arms: Patients undergoing upper gastrointestinal endoscopy with head box

SUMMARY:
According to preexisting data, it has revealed the fundamental role that aerosols play in the transmission of the COVID-19 virus. Esophagogastroduodenoscopy (EGD), producing particle smaller than 5 microns, was regarded as 'aerosol-generating procedures' (AGPs) associated with an increased risk of transmission of respiratory pathogens to healthcare workers. The strategies aim to reduce spreading of aerosol during the procedure should be beneficial. Using an acrylic box to cover the head of a patient undergoing an endoscopy seems to reduce aerosol scatter and reduce the spread of respiratory pathogens. At present, there are no high-quality studies that provide quantitative data on the use of head box to reduce aerosol generation.

DETAILED DESCRIPTION:
Pandemic of coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) affected globally clinical practice including temporary postponement of elective endoscopic procedures in GI office activity and has caused an unprecedent concern in personal protection against the airborne virus. Whitin 2.5 years since the outbreak in mid-December 2019, COVID-19 had infected over 182 million people and killed more than 3.9 million across 210 countries worldwide. (Ref. https://www.who.int/emergencies/diseases/novel-coronavirus-2019).

According to preexisting data, it has revealed the fundamental role that aerosols play in the transmission of the COVID-19 virus. Previously, in the medical community attempted to find strategies to minimize risk of respiratory transmission to HCPs during pandemic such as wearing either standard or full personal protective equipment (PPE), including do-it-yourself devices and gadgets are the necessary substitutes to protect them from aerosolization. However, there has been no published study evaluating the efficacy or real benefit of these tools in preventing aerosolization during EGD quantitatively.

Esophagogastroduodenoscopy (EGD), producing particle smaller than 5 microns, was regarded as 'aerosol-generating procedures' (AGPs) associated with an increased risk of transmission of respiratory pathogens to healthcare workers. The strategies aim to reduce spreading of aerosol during the procedure should be beneficial.

Using an acrylic box to cover the head of a patient undergoing an endoscopy seems to reduce aerosol scatter and reduce the spread of respiratory pathogens. At present, there are no high-quality studies that provide quantitative data on the use of head box to reduce aerosol generation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who indicated in upper gastrointestinal endoscopy and undergoing endoscopy at Excellence Center For GI Endoscopy, King Chulalongkorn Memorial Hospital, Thailand
* Age of 18 years or more

Exclusion Criteria:

* Patients with a high risk of conscious sedation who need an anesthetist
* Patients with refusal to participate in clinical research
* Patients who cannot make medical decisions on their own
* Patients who underwent therapeutic endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The amount of aerosol particles measured on the face of th endoscopist performing an upper gastrointestinal endoscopy | 5 months
  Aerosol particles measured by portable particle counter as count per cubic foot

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meselson M. Droplets and Aerosols in the Transmission of SARS-CoV-2. N Engl J Med. 2020 May 21;382(21):2063. doi: 10.1056/NEJMc2009324. Epub 2020 Apr 15. No abstract available. PMID 32294374
- [Result] Hennessy B, Vicari J, Bernstein B, Chapman F, Khaykis I, Littenberg G, Robbins D. Guidance for resuming GI endoscopy and practice operations after the COVID-19 pandemic. Gastrointest Endosc. 2020 Sep;92(3):743-747.e1. doi: 10.1016/j.gie.2020.05.006. Epub 2020 May 11. No abstract available. PMID 32437712
- [Result] Yu IT, Li Y, Wong TW, Tam W, Chan AT, Lee JH, Leung DY, Ho T. Evidence of airborne transmission of the severe acute respiratory syndrome virus. N Engl J Med. 2004 Apr 22;350(17):1731-9. doi: 10.1056/NEJMoa032867. PMID 15102999
- [Result] Somsen GA, van Rijn CJM, Kooij S, Bem RA, Bonn D. Measurement of small droplet aerosol concentrations in public spaces using handheld particle counters. Phys Fluids (1994). 2020 Dec 1;32(12):121707. doi: 10.1063/5.0035701. PMID 33362399
- [Result] Chan SM, Ma TW, Chong MK, Chan DL, Ng EKW, Chiu PWY. A Proof of Concept Study: Esophagogastroduodenoscopy Is an Aerosol-Generating Procedure and Continuous Oral Suction During the Procedure Reduces the Amount of Aerosol Generated. Gastroenterology. 2020 Nov;159(5):1949-1951.e4. doi: 10.1053/j.gastro.2020.07.002. Epub 2020 Jul 7. No abstract available. PMID 32649933
- [Result] Sagami R, Nishikiori H, Sato T, Tsuji H, Ono M, Togo K, Fukuda K, Okamoto K, Ogawa R, Mizukami K, Okimoto T, Kodama M, Amano Y, Murakami K. Aerosols Produced by Upper Gastrointestinal Endoscopy: A Quantitative Evaluation. Am J Gastroenterol. 2021 Jan 1;116(1):202-205. doi: 10.14309/ajg.0000000000000983. PMID 33079747
- [Result] Gregson FKA, Shrimpton AJ, Hamilton F, Cook TM, Reid JP, Pickering AE, Pournaras DJ, Bzdek BR, Brown J; AERATOR group. Identification of the source events for aerosol generation during oesophago-gastro-duodenoscopy. Gut. 2022 May;71(5):871-878. doi: 10.1136/gutjnl-2021-324588. Epub 2021 Jun 29. PMID 34187844
- [Result] Pittayanon R, Faknak N, Ananchuensook P, Prasoppokakorn T, Plai-Dum S, Thummongkhol T, Paitoonpong L, Rerknimitr R. Amount of contamination on the face shield of endoscopists during upper endoscopy between patients in two positions: A randomized study. J Gastroenterol Hepatol. 2021 Jul;36(7):1913-1919. doi: 10.1111/jgh.15416. Epub 2021 Feb 18. PMID 33506983